CLINICAL TRIAL: NCT06960512
Title: The Impact of Precision Lifestyle Intervention on Blood Glucose Control in Type 2 Diabetes Mellitus
Brief Title: Precision Lifestyle Interventions Guided by Continuous Glucose Monitoring: Impact on Glycemic Outcomes in Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QTK 2025-0001
Record Dates: First submitted 2025-04-26; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: lifestyle medicine; Type 2 Diabetes Mellitus; continuous glucose monitoring; HBA1c; Glycosylated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision Lifestyle Intervention (PLI) group (Experimental)
  Interventions: Behavioral: Precision Lifestyle Intervention (PLI) group
- Health Education (HE) group (No Intervention)

INTERVENTIONS:
Behavioral: Precision Lifestyle Intervention (PLI) group — 1. Device Application: Participants in the intervention group will wear the GX-01S continuous glucose monitoring system, with data transmitted in real-time to a secure cloud platform.
  2. Multidisciplinary Management: A specialized team (health managers, nutritionists, endocrinologists, and Counselor) will analyze glucose fluctuations, dietary patterns, sleep health, physical activity and to formulate personalized adjustment plans. Modifications may include meal timing optimization, sleep duration regulation, and exercise frequency adaptations.
  3. Telehealth Follow-up: Participants will receive structured guidance via telephone/telemedicine consultations throughout the 28-day intervention period. Type 2 Diabetes Mellitus (T2DM) patient compliance will be systematically monitored and documented.
  4. Tailored Recommendations: Evidence-based lifestyle recommendations will be provided post-intervention, informed by quantitative biomarker data and adherence metrics collected.
  Arms: Precision Lifestyle Intervention (PLI) group

SUMMARY:
This study is an interventional research. Through scientific evaluation, it explores the effect of precise lifestyle intervention based on CGM data on the control of chronic type 2 diabetes mellitus. By formulating a safe and effective precise lifestyle intervention plan, lifestyle medicine is integrated into the management of chronic diseases. Through multidimensional evaluations, it is expected to improve patients' self-management ability and provide a reference for the development of chronic diabetes management.

DETAILED DESCRIPTION:
Internationally, significant breakthroughs have been made in diabetes research. The 'Standards of Care in Diabetes-2024' released by the ADA has shifted treatment goals from solely lowering blood glucose to comprehensive control of blood sugar, protecting target organs, reducing complications, and improving the overall prognosis for diabetes patients. It also emphasizes the importance of medical care providers mastering new technologies, such as using artificial intelligence for retinal screening and making necessary referrals, adopting telemedicine and digital tools for diabetes self-management education, personalized guidance, and the chronic disease management model is increasingly maturing. In China, diabetes management models include hospital management, community management,'hospital-community integration', and information technology-assisted management, etc. They face issues such as inconsistent standards and low efficiency. At the same time, they tend to focus more on the control of physical and chemical indicators, while lacking sufficient attention to the related symptoms, quality of life, and psychological state of diabetes patients.

This study is an interventional research.With the main purpose of 'exploring the impact of precise lifestyle interventions based on CGM data on blood glucose control in T2DM patients', this study aims to scientifically evaluate the effects of precise lifestyle interventions based on CGM data on chronic disease control in type2 diabetes diabetes mellitus. By formulating a safe and effective precise lifestyle intervention plan, lifestyle medicine is integrated into the management of chronic diseases. Through multidimensional evaluations, such as target management, lifestyle intervention, dietary intervention, exercise therapy, mental health, monitoring of diabetes-susceptible genes, and intervention of gut microbiota gene detection, it is expected to improve patients' self-management ability and provide a reference for the development of chronic diabetes management.

The purpose is to enhance patients' self-management capabilities, improve the quality of primary healthcare services, assist medical staff in developing and refining personalized treatment plans, reduce the incidence of diabetes complications, enhance patients' quality of life and life expectancy, promote scientific progress in the field of diabetes management, and effectively address the challenges of chronic diseases in an aging society.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the diagnostic criteria for T2DM in the 'Clinical guidelines for prevention and treatment of type 2 diabetes mellitus in the elderly in China (2020 edition)', and be diagnosed with type 2 diabetes mellitus, i.e., mainly due to insulin resistance and insufficient relative insulin secretion, and have the typical symptoms of diabetes mellitus (irritable thirst and excessive drinking, excessive urination, excessive food intake, and unexplained weight loss) plus a random glucose level ≥11.1 mmol/L (200 mg/dl), or plus a fasting Blood glucose level ≥ 7.0 mmol/L (126 mg/dl), or plus random blood glucose or OGTT (Oral Glucose Tolerance Test) 2-hour blood glucose level ≥ 11.1 mmol/L (200 mg/dl), or plus glycated hemoglobin (HbA1c) level ≥ 6.5%;
* Age 18～65 years old (including the threshold), gender is not limited;
* Can skillfully operate a smartphone by themselves, or their family members can help to use the phone to give feedback on their daily life situation;
* Willing to participate in this study with good compliance;
* Agree to authorize He Eye Specialist Hospital to make cases of health management content.

Exclusion Criteria:

* Pregnant women, lactating women, and women of childbearing age who do not wish to use contraception during the research period;
* Severe skin disease, adhesive tape or adhesive allergy at the sensor placement site;
* People with a history of specific allergies, or allergies (e.g., allergic to two or more drugs, food, or pollen);
* Patients who meet the criteria for Grade 3 hypertension according to the ratings in the' Chinese Guidelines for the Prevention and Treatment of Hypertension (2024 Revision)', i.e., blood pressure over 180/110 mmHg, or low blood pressure of 110 mmHg or more;
* Suffering from severe cardiovascular and cerebrovascular diseases (including ST-segment elevation myocardial infarction, unstable angina up to Braunwald classification III (one or more episodes of resting angina within 48 hours), transient ischemic attack, stroke treatment accompanied by various degrees of sequelae (e.g.,hemiplegia,aphasia,impaired consciousness, epilepsy, and even dementia), coronary artery stenosis of moderate stenosis (50%) and above, hemodialysis reconstruction surgery less than 6 months, cerebral embolism and cerebral hemorrhage less than 6 months or with varying degrees of movement disorders after the treatment, cognitive disorders, speech and swallowing disorders, and other sequelae, etc.), or daily accompanied by frequent episodes of angina pectoris, chest tightness, chest pain and other symptoms;
* Renal insufficiency up to stage III and above (blood creatinine level more than 450μmol/L);
* History of psychoSsis or psychotropic substance abuse;
* Any condition judged by the investigator to be unsuitable for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin/ HbA1c | Time Frame:On the 0th, 28th, and 90th days of the trial.
  It reflects average blood glucose levels over the past 2-3 months and is used to diagnose and monitor diabetes management and will be done 3 times at every assessment session and the median value will be recorded.
fasting blood glucose/FBG | Time Frame:On the 0th, 28th, and 90th days of the trial.
  Fasting blood glucose measures blood sugar levels after an 8-hour fast and is primarily used to diagnose diabetes or prediabetes. The measurements will be done 3 times at every assessment session and the median value will be recorded.

SECONDARY OUTCOMES:
Total Cholesterol/TC | Time Frame:On the 0th, 28th, and 90th days of the trial.
  TC (Total Cholesterol) measures the total concentration of cholesterol in the blood, including LDL, HDL, and triglycerides, and is used to evaluate cardiovascular health, lipid metabolism status and guide lipid management.
Triglycerides/TG | Time Frame:On the 0th, 28th, and 90th days of the trial.
  TG (Triglycerides) measures the level of triglycerides in the blood and is used to evaluate cardiovascular risk, metabolic disorders, or abnormalities in lipid metabolism.
Blood Pressure/BP | Time Frame:On the 0th, 28th, and 90th days of the trial.
  BP (Blood Pressure)measures the pressure exerted by blood on arterial walls during heart contractions (systolic) and relaxations (diastolic), and is used to assess cardiovascular health, hypertension, or hypotension.
urinalysis/UA | Time Frame:On the 0th, 28th, and 90th days of the trial.
  A urinalysis analyzes the physical, chemical, and microscopic properties of a urine sample to detect abnormalities and help diagnose conditions such as urinary tract infections, kidney disorders, or metabolic diseases.
Diabetic Retinopathy Screening (DRS) via Fundus Photography | Time Frame:On the 0th, 28th, and 90th days of the trial.
  Fundus photography is a non-invasive imaging method that captures high-resolution images of the retina, optic disc, and blood vessels. It is utilized to evaluate the presence and severity of diabetic retinopathy (e.g., microaneurysms, hemorrhages, neovascularization) and monitor diabetes-related ocular complications.The assessment will be performed once at each session, with results documented for analysis.Retinal Image Biomarker Analysis is about to get digits like Retinal vessel diameter,Retinal vessel tortuosity,Retinal vascular fractal dimension,Retinal vessel bifurcation patterns, etc.These microvascular metrics will be analyzed to evaluate diabetes-induced alterations in retinal microcirculation, providing objective biomarkers for early microvascular dysfunction and disease progression monitoring. All parameters will be measured using validated automated image analysis software.

IPD SHARING:
Plan to Share IPD: No